CLINICAL TRIAL: NCT03289312
Title: Dissecting How Peripheral Lymphocytes Are Lost During Sepsis
Acronym: SLL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jianfeng Xie, Southeast University, China, Southeast University, China
Other Study IDs: 2017ZDSYSLLoss
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Last update posted 2017-12-27 (Actual); Status verified 2017-09

CONDITIONS: Sepsis
Keywords: sepsis, lymphocyte
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sepsis: Diagnosis of new onset sepsis within 24h without history of tumor, hematological or immunological disease, and treatment with chemotherapy agents or corticosteroids within 6 months prior to or during the hospitalization.
- Health control: Health vonlunteers

SUMMARY:
There is an observational, clinical study. We recruit sepsis patients to investigate what drives peripheral lymphocyte loss in sepsis.

DETAILED DESCRIPTION:
There is an observational, clinical study. We recruit patients with diagnosis of new onset sepsis within 24h, collect and record clinical characteristics：

①Demography data，diagnosis, admission source, infection source, APACHE II,SOFA scores;②Endotoxin levels and PaO2 measured;③Immune and systemic inflammatory indicators：T, RR, WBC, ALC, etc.;④Complicated organs dysfunctions: duration and therapy;⑤Incidence of ICU-acquired infection and prognosis.The blood samples were collected for apoptosis,necrosis,autophagy,pyroptosis measurements.The aim of this study is to investigate how peripheal lymphocyte loss relates to outcome and the mechanisms of peripheal lymphocyte loss in different condition.

ELIGIBILITY:
Inclusion Criteria:

* Health volunteers

Exclusion Criteria:

* History of tumor, hematological or immunological disease, and treatment with chemotherapy agents or corticosteroids within 6 months prior to or during the hospitalization.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  * Diagnosis of new onset sepsis within 24h.
  Exclusion Criteria:
  * History of tumor, hematological or immunological disease, and treatment with chemotherapy agents or corticosteroids within 6 months prior to or during the hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2018-01-11 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
lymphocyte loss | day of inclussion and 7th day after inclussion
  ratios of T cells loss by different mechanism in different subgroups

SECONDARY OUTCOMES:
prognosis | 28-day after inclussion
  28-day prognosis:survive or not
Complicated organ dysfunction | during 28 days after inclussion
  duration and surpport therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided